CLINICAL TRIAL: NCT03927404
Title: Development of Adaptive Vacuum Suspension to Improve Prosthetic Fit and Residual Limb Health
Acronym: DoD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Chandan Sen, Associate Vice President of Research, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1809327674; W81XWH-16-2-0059 (Other Grant/Funding Number: DoD)
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Lower Limb Amputation
Keywords: Transfemoral Amputees; Transtibial Amputees; Prosthesis

STUDY DESIGN:
Intervention Model Description: This is a 16 weeks longitudinal study where subjects will serve their own control. A baseline measurement will be done prior to start of intervention that will continue for 16 weeks and a final measurement will be taken at the end of 16 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Adaptive Vacuum test Prosthesis (Experimental): The experimental socket system uses an active vacuum pump to push air out of the socket. The level of vacuum is controlled by hardware that automatically detects the socket fit based on in-socket motion and adjusts vacuum as needed to eliminate this motion.
  Interventions: Device: Active vacuum test prosthesis

INTERVENTIONS:
Device: Active vacuum test prosthesis — The adaptive vacuum prosthesis is sold as a commercial device by the company Willow Wood with suggested U.S. L-Code L5781. The device is designated as a Class 1 Medical Device and 510(K) Exempt. This category is part of a low or moderate risk to patient safety and health. The Prosthetic socket system uses an active vacuum pump to push air out of the socket. The level of vacuum is controlled by hardware that automatically detects the socket fit based on in-socket motion and adjusts vacuum as needed to eliminate this motion.
  Other Names: Limb logic system

SUMMARY:
The purpose of the study is to evaluate residual limb circulation and skin health associated with the use of a prosthetic vacuum socket. A conventional non-vacuum prosthetic socket will be compared to a vacuum prosthetic socket.

The prosthetic suspension plays a pivotal role in an amputee's comfort. It can also significantly impact an amputee's limb health. If the prosthesis is not held securely to the amputee's limb, relative movement between the limb and prosthetic interface can cause bruising, skin irritation and skin breakdown. These poor outcomes are uncomfortable and can lead to much more serious health conditions. A positive solution to creating secure and comfortable suspension is the use of a vacuum suspension socket. The vacuum pressure assists in preventing movement in the socket. The clinical benefits associated with vacuum suspension include volume retention, increased proprioception, secure suspension, and frequently reported observations of wound healing. However, the long term effects of vacuum suspension on circulation remain undetermined or undocumented. This study examines a vacuum suspension system on the health of the residual limb (amputated limb). A vacuum socket creates a vacuum between the rigid prosthetic socket and prosthetic liner which is sealed to the socket. Therefore, vacuum is not directly applied to the skin of the residual limb.

DETAILED DESCRIPTION:
There are a total of 3 study visits, (some visits may be broken into separate visits per preference of subject), including socket fitting visits (which could be 2 separate visits), a baseline visit, and a final visit. During the socket visit, which may consist of a three visits plus socket adjustments (as needed by the participant) on separate days (up to 4 weeks), limb shape capture, measurement or tracing, diagnostic static fitting and diagnostic static fitting, and delivery of a definitive "research" socket will be done. At the baseline visit, participants will perform seated tasks, standing tasks, and treadmill walking tasks. Residual limb health measurements will be taken before and after the activity period, including surface electrical capacitance, Transepidermal Water Loss (TEWL) measurement, hyperspectral imaging, Hitachi Aloka ultrasound imaging, Blood Flow, and digital imaging during the baseline visit as well. The final visit, using the research socket, will consist of the same tasks and measurements as the baseline visit and questionnaires will be completed. The subject may choose to break up the final visit tasks into 2 different visits if desired.

After completion of the study, participants will be given the choice to keep the research socket or return to using their original prosthesis as normal. The study prosthetist will be available to review and adjust the fit of their standard of care prosthesis at this time. Note: Due to physical change and limb volume fluctuation over the study period, it is possible that at the end of the study the standard of care prosthesis will not fit your residual limb as it does at the beginning of the study. At the completion of the study, it is recommended that the subject follow up with their primary care prosthetist for socket evaluation and fitting.

There may be risks that are not known about at this time. Side effects, risks, and discomforts may result from study participation .While the goal of this project is to create a more comfortable prosthesis, it is possible that the subject could experience discomforts commonly associated with prosthesis use, such as perspiration, dry skin, rash, itching, blisters, high pressure in the socket, looseness in the socket, and mechanical rubbing that leads to ulceration which may lead to infection and additional surgery. Subjects with low levels of arterial blood flow have an additional risk of ulceration.

* Prosthesis placement: While the goal of this project is to create a more comfortable prosthesis, it is possible that the subject could experience discomforts commonly associated with prosthesis use, such as perspiration, dry skin, rash, itching, blisters, high pressure in the socket, looseness in the socket, and mechanical rubbing that leads to ulceration.
* Treadmill task:There is a risk of falling during the research activities. This risk is mitigated by the ability of participants to self-select pace for the treadmill task and observation of treadmill activities by research staff.
* Transcutaneous Oxygen Measurement (TcOM) and skin temperature: The PeriFlux System 5000 uses non-invasive probes that will measure the skin temperature and transcutaneous Oxygen Measurement and poses minimal risk to the subject. The probe head is affixed to the residual limb by an adhesive sticker. Removal of the sticker after data acquisition may cause minor discomfort similar to removing a small band-aid.
* Hyperspectral Imaging: This non-invasive imaging technique poses minimal risk to the subject. A small fiduciary marker sticker is placed on the subject's limb to calibrate camera settings. Removal of the sticker after imaging may cause minor discomfort similar to removing a small band-aid.
* Hitachi Aloka Ultrasound:Ultrasound imaging is a noninvasive technique and is a minimal risk procedure.
* TEWL and Surface Electrical Capacitance Measurements: TEWL and Surface Electrical Capacitance measurements are noninvasive and propose less than minimal risk.

Subjects will be queried on self-reported measures of user comfort and performance. Briefly, four subjective measures will be completed: VR-36, PEQ, SCS, and measures from the NIH PROMIS

The CHAMP test will be used to assess overall amputee performance and the effect of the socket suspension intervention over time. The conglomeration of clinical assessment tools into the CHAMP was specifically done to measure high-level mobility in service members with a lower limb amputation. CHAMP consists of the Single Leg Stance Test (SLS), the Edgren Side Step Test (ESST), Illinois Agility Test (IAT), and T Test.

IU Neuroscience Gait lab will be used to collect kinematic data. The laboratory is equipped with an instrumented treadmill and infrared camera system. A harness system will be used to provide support and safety for the amputees while study participants walk on the treadmill for 6 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18 and above
* Unilateral transtibial or transfemoral amputee
* Ambulate at a K2 level or higher
* At least 3 months post-amputation per physician discretion
* Residual limb length greater than 6.5 inches in length
* Able to follow directions and give informed consent on their own or through Legally Authorized Representative.
* Must be able to ambulate without assistance. An external assistance device such as cane or walker will be permitted.
* Adequate arterial blood flow as evidenced by a TcOM >30mmHg measured within the past 12 months.

Exclusion Criteria:

* Conditions that prevent wearing a prosthetic socket,such as existing scab, ulcer, or keloid scar on amputation stump.
* Cognitive deficits or mental health problems that would limit ability to consent and participate fully in the study protocol
* Women who are pregnant or who plan to become pregnant in the near future

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandan Sen, PhD, Principal Investigator — Indiana University
Locations (1):
- IU Health Methodist Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Epstein RA, Heinemann AW, McFarland LV. Quality of life for veterans and servicemembers with major traumatic limb loss from Vietnam and OIF/OEF conflicts. J Rehabil Res Dev. 2010;47(4):373-85. doi: 10.1682/jrrd.2009.03.0023. PMID 20803405
- [Background] Schultz AE, Baade SP, Kuiken TA. Expert opinions on success factors for upper-limb prostheses. J Rehabil Res Dev. 2007;44(4):483-9. doi: 10.1682/jrrd.2006.08.0087. PMID 18247245
- [Background] Zachariah SG, Saxena R, Fergason JR, Sanders JE. Shape and volume change in the transtibial residuum over the short term: preliminary investigation of six subjects. J Rehabil Res Dev. 2004 Sep;41(5):683-94. doi: 10.1682/jrrd.2003.10.0153. PMID 15558398
- [Background] Fernie GR, Holliday PJ. Volume fluctuations in the residual limbs of lower limb amputees. Arch Phys Med Rehabil. 1982 Apr;63(4):162-5. PMID 7082139
- [Background] Sanders JE, Fatone S. Residual limb volume change: systematic review of measurement and management. J Rehabil Res Dev. 2011;48(8):949-86. doi: 10.1682/jrrd.2010.09.0189. PMID 22068373
- [Background] Krueger CA, Wenke JC, Ficke JR. Ten years at war: comprehensive analysis of amputation trends. J Trauma Acute Care Surg. 2012 Dec;73(6 Suppl 5):S438-44. doi: 10.1097/TA.0b013e318275469c. PMID 23192067
- [Background] Ramasamy A, Hill AM, Phillip R, Gibb I, Bull AM, Clasper JC. The modern "deck-slap" injury--calcaneal blast fractures from vehicle explosions. J Trauma. 2011 Dec;71(6):1694-8. doi: 10.1097/TA.0b013e318227a999. PMID 21808204
- [Background] Bui KM, Raugi GJ, Nguyen VQ, Reiber GE. Skin problems in individuals with lower-limb loss: literature review and proposed classification system. J Rehabil Res Dev. 2009;46(9):1085-90. doi: 10.1682/jrrd.2009.04.0052. PMID 20437314
- [Background] Harris AM, Althausen PL, Kellam J, Bosse MJ, Castillo R; Lower Extremity Assessment Project (LEAP) Study Group. Complications following limb-threatening lower extremity trauma. J Orthop Trauma. 2009 Jan;23(1):1-6. doi: 10.1097/BOT.0b013e31818e43dd. PMID 19104297

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were enrolled at CWC Methodist Indiana University Health and Willow Wood Ohio
Pre-assignment Details: any subject did not meet the blood perfusion eligibility criteria were screened failed
Groups:
- Adaptive Vacuum Test Prosthesis: This is a crossover study design where participant come in their standard of care socket suspension system and the baseline measurements are performed followed by a 16 week period in the experimental socket system that uses an active vacuum pump to push air out of the socket. The level of vacuum is controlled by hardware that automatically detects the socket fit based on in-socket motion and adjusts vacuum as needed to eliminate this motion.
  Active vacuum test prosthesis: The adaptive vacuum prosthesis is sold as a commercial device by the company Willow Wood with suggested U.S. L-Code L5781. The device is designated as a Class 1 Medical Device and 510(K) Exempt. This category is part of a low or moderate risk to patient safety and health. The Prosthetic socket system uses an active vacuum pump to push air out of the socket. The level of vacuum is controlled by hardware that automatically detects the socket fit based on in-socket motion and adjusts vacuum as needed to eliminate this motion.
Period: Overall Study
Arm/Group | Adaptive Vacuum Test Prosthesis
Started (Primary outcomes are measured in their Standard of care socket system as baseline value followed by initiation of using the test socket for 16 weeks.) | 60
Completed | 59
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adaptive Vacuum Test Prosthesis
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 59
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 47
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59
Age [Median (Inter-Quartile Range); unit: years] | 57 [39 to 63]

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Trans-epidermal Water Loss (TEWL) at 16 Weeks After Use
Description: Trans-epidermal Water Loss in 16 wks. Higher TEWL value represents a worse outcome with loss of skin barrier function.
  The value reported is the ratio of the TEWL of residual limb over TEWL value of the sound side limb.
Time Frame: Baseline and 16 Weeks
Population: A total of n=60 subjects were enrolled at IU (n=30) and WW (n=30) sites. One enrolled subject discontinued and therefore n=59 subjects were analyzed. The studies initiated mid-2019, however, due to global pandemic research activities were greatly affected at both sites. The studies were on hold and got reinitiated fall of 2020 at IU and WW sites. Declaration of Helsinki protocols was followed, and patients gave their written informed consent.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Adaptive Vacuum Test Prosthesis
Number analyzed (Participants) | 59
ratio | 1.69 [1.12 to 2.85]
Statistical Analysis 1: Comparison: Adaptive Vacuum Test Prosthesis; Test type: Other — We used median (Inter-quartile range) to describe the continuous measures of limb health such as TEWL, Hydration, and Oxygenation levels at each visit and each location of the measurements in the sound (SL) and residual limbs (RL); p < 0.05, bivariate analysis — In a bivariate analysis, we used two-sided equality of the median test for the matched pairs of observations

2. Secondary Outcome: Change in Hyperspectral Imaging at 16 Wks
Description: Change from baseline in Hyperspectral Imaging at 16 wks; tissue oxygenation measured using hyperspectral imaging. Higher the HbO2 better is the perfusion in skin indicating less damage.
Time Frame: Baseline to16 weeks
Population: total of n=60 subjects were enrolled at IU (n=30) and WW (n=30) sites. One enrolled subject discontinued and therefore n=59 subjects were analyzed. The studies initiated mid-2019, however, due to global pandemic research activities were greatly affected at both sites. The studies were on hold and got reinitiated fall of 2020 at IU and WW sites. Declaration of Helsinki protocols was followed, and patients gave their written informed consent.
Measure: Median (Inter-Quartile Range); unit: Percentage of Oxygen
Arm/Group | Adaptive Vacuum Test Prosthesis
Number analyzed (Participants) | 59
Percentage of Oxygen | 1.2 [0.55 to 2.94]

3. Secondary Outcome: Ultrasound Measurements at 16 Wks
Description: In elasto-mode the blue color represents less elastic skin and weak tensile strength. whereas red is more elastic skin and high tensile strength. The blue & red color intensities in elasto mode were calculated in Matlab as arbitrary units (AU). The data presented is median of the AU. A lower AU meaning better tensile strength of the tissue meaning favorable outcome.
Time Frame: 16 weeks
Population: A total of n=60 subjects were enrolled at IU (n=30) and WW (n=30) sites. The data that passed QC for the analysis was n=23 used for final data.
Measure: Median (Inter-Quartile Range); unit: Arbitrary Units (AU)
Arm/Group | Adaptive Vacuum Test Prosthesis
Number analyzed (Participants) | 23
Arbitrary Units (AU) | 1.2508 [0.856 to 1.88]
Statistical Analysis 1: Comparison: Adaptive Vacuum Test Prosthesis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.05, bivariate analysis — In a bivariate analysis, we used two-sided equality of the median test for the matched pairs of observations

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: same as Ct.gov definitions
Arm/Group | Adaptive Vacuum Test Prosthesis
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT03927404/Prot_SAP_003.pdf